CLINICAL TRIAL: NCT06172933
Title: A Text- and Audio-based Intervention to Promote Physical Activity in Midlife
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Celano, Associate Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P003312
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Middle Aged
Keywords: Text message; Podcast; Well-being; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, wait-list controlled, blinded intervention trial
Who Masked: Outcomes Assessor
Masking Description: While participants and study trainers will be aware of group assignment, a blinded study team member will perform outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Move with Meaning (Experimental): In Move with Meaning, participants will engage in twice weekly, interactive text message sessions, which are accompanied by audio content to promote engagement in the program. In the first session of each week, participants will review their physical activity goal and positive psychology topic from last week, then learn about a new positive psychology and physical activity topic and ultimately set a new physical activity goal for the week. In the second session, participants will either be reminded of the content of the audio file and the goal they set earlier that week. The program will run for eight weeks.
  Interventions: Behavioral: Move with Meaning
- Wait-list control (No Intervention): Participants in the wait-list control condition will engage in usual medical care for eight weeks, then will complete the Move with Meaning program.

INTERVENTIONS:
Behavioral: Move with Meaning — Participants will engage in twice weekly text message sessions, will listen to a weekly audio session, and will work towards a physical activity goal each week, for a total of eight weeks.
  Arms: Move with Meaning

SUMMARY:
This is a randomized, controlled pilot trial (N=30) to examine the feasibility, acceptability, and preliminary efficacy of the Move with Meaning program, an 8- week, text message- and audio-based intervention to promote physical activity in midlife adults.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot trial to examine the feasibility, acceptability, and preliminary efficacy of the Move with Meaning program, an 8- week, text message- and audio-based intervention to promote physical activity in midlife adults. In Move with Meaning, participants will listen to weekly audio sessions and complete twice weekly text message sessions, in which they will set a weekly physical activity goal. The primary outcome is feasibility (measured by number of successful text message sessions sent). Secondary outcomes include acceptability and preliminary impact on physical activity, psychological health-, and physical health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Midlife adults (aged 45-64 years at the time of enrollment)
* Suboptimal physical activity (<150 minutes of moderate to vigorous physical activity, measured by accelerometer)
* Access to a phone capable of receiving text messages and listening to audio files (i.e., a smartphone)

Exclusion Criteria:

* An unrelated condition limiting physical activity
* Participation in any other programs focused on cardiac prevention or well-being
* A cognitive disturbance precluding participation or informed consent
* Current pregnancy
* Inability to speak/write fluently in English

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of text message sessions successfully delivered | Weekly over 8 weeks
  The automated platform will record rates of successful text message delivery.

SECONDARY OUTCOMES:
Proportion of audio sessions completed by participants | Weekly over 8 weeks
  We will record the number of sessions in which participants engaged (e.g., responded to a text message), out of a total of 8 sessions.
Session utility | Weekly over 8 weeks
  Participants will rate the utility of each session, measured on a 10-point Likert scale. Higher scores indicate greater utility.
Change in overall physical activity (in steps/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  Physical activity (steps) will be measured via an Actigraph accelerometer. We will use established accelerometer protocols to measure the mean number of steps taken per day at each time point.
Change in moderate to vigorous physical activity (MVPA; in mean minutes/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  MVPA (reported in mean minutes of MVPA/day) will be measured via an Actigraph accelerometer and recorded in mean minutes/day.
Change in sedentary time (in mean minutes/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  Sedentary time (mean minutes/day) will be measured via Actigraph accelerometer.
Change in self-reported physical activity (International Physical Activity Questionnaire [IPAQ]; in metabolic equivalent-minutes/week) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  This will be measured via the International Physical Activity Questionnaire (IPAQ) as a secondary measure of physical activity.
Change in positive affect (Positive and Negative Affect Schedule [PANAS] positive affect items) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Positive affect (our main psychological outcome given its links to health outcomes and sensitivity to change) will be assessed via the Positive and Negative Affect Schedule (PANAS) positive affect items. PANAS scores range from 10-50, with higher scores indicating higher levels of positive affect.
Change in optimism (Life Orientation Test - Revised [LOT-R]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Optimism will be measured using the Life Orientation Test - Revised (LOT-R), a frequently used 6-item instrument that assesses dispositional optimism. LOT-R scores range from 0-24, with higher scores indicating higher levels of optimism.
Change in depressive symptoms (depression subscale of the Hospital Anxiety and Depression Scale [HADS]). | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Depressive symptoms will be measured using the 7-item depression subscale of the Hospital Anxiety and Depression Scale (HADS). The depression subscale of the HADS ranges from 0-21, with higher scores indicating higher levels of depression.
Change in anxiety (anxiety subscale of the Hospital Anxiety and Depression Scale [HADS]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Anxiety will be measured using the 7-item anxiety subscale of the Hospital Anxiety and Depression Scale (HADS). The anxiety subscale of the HADS ranges from 0-21, with higher scores indicating higher levels of anxiety.
Change in exercise self-efficacy (Self-Efficacy for Exercise scale [SEE]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Exercise self-efficacy will be measured via the Self-Efficacy for Exercise (SEE) scale. SEE scores range from 0-90, with higher scores indicating higher levels of self-efficacy for exercise.
Change in perceived social support (Multidimensional Scale of Perceived Social Support) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Perceived social support will be measured by the Multidimensional Scale of Perceived Social Support (MSPSS). MSPSS scores range from 1-7, with higher scores indicating higher levels of perceived social support.
Change in internal health locus of control (Multidimensional Health Locus of Control [MHLC] scale) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Internal locus/sense of control will be measured using the Multidimensional Health Locus of Control (MHLC) scale. The internal locus of control score from the MHLC ranges from 6-36, with higher scores indicating greater internal locus of control.
Change in positive affect during activity (Physical Activity Enjoyment Scale) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Positive affect during activity will be measured using the Physical Activity Enjoyment Scale. Physical Activity Enjoyment Scale scores range from 18-126, with higher scores indicating higher levels of enjoyment during activity.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No